CLINICAL TRIAL: NCT01320800
Title: CBT for Social Anxiety Disorder Delivered by School Counselors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MH81881; R01MH081881 (NIH); NCT01892735 (obsolete NCT alias)
Record Dates: First submitted 2011-03-11; First posted 2011-03-22 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Expert-led CBT (Active Comparator): Expert SASS is the Skills for Academic and Social Success protocol delivered by a postdoctoral fellows.
  Interventions: Behavioral: Skills for Academic and Social Success
- School Counselor-led CBT (Experimental): School Counselor SASS is the Skills for Academic and Social Success protocol delivered by School Counselors.
  Intervention: Behavioral: Skills for Social and Academic Success
  Interventions: Behavioral: Skills for Academic and Social Success
- Skills for Life (Active Comparator): SFL is the Skills for Life Protocol delivered by school counselors. Intervention: Behavioral: Skills for Life
  Interventions: Behavioral: Skills for Life

INTERVENTIONS:
Behavioral: Skills for Academic and Social Success — 12-week cognitive-behavioral, school-based group intervention
  Arms: Expert-led CBT; School Counselor-led CBT
Behavioral: Skills for Life — SFL is the Skills for Life Protocol delivered by school counselors.
  Arms: Skills for Life

SUMMARY:
This 5-year study addresses the unmet needs of adolescents with social phobia through the testing of a 12-week cognitive-behavioral, school-based group intervention delivered by trained school counselors compared to a nonspecific school counseling program. A secondary goal is to provide further examination of the efficacy of the CBT program delivered by school counselors as compared to the same program delivered by psychologists.

DETAILED DESCRIPTION:
The investigators have tested SASS, a school-based group CBT intervention for social phobia, and found it to be effective when delivered by psychologists (Masia Warner et al., 2005; Masia Warner et al., 2007). The proposed dissemination study extends this work through a controlled trial of SASS delivered by school counselors. The investigators will randomize 126 adolescents with social anxiety disorder, ages 14 through 17, to one of 3 treatments: 1) SASS delivered by school counselors (SC-SASS), 2) SASS delivered by psychologists (Expert-SASS), or 3) a manualized adolescent group counseling program specifically designed for school counselors, called Skills for Living (SFL). A comprehensive evaluation will include diagnosis, illness severity, scale ratings of social anxiety and depression, clinical global improvement, overall functioning, and school-relevant indices of function. Outcomes will be assessed at baseline, mid-point (after 6 weeks of intervention), post-treatment, and 6 months following intervention completion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis. DSM-IV primary diagnosis (most severe) of social anxiety disorder (as determined by the ADIS-PC)
2. Age and Sex. Boys and Girls, 14 through 19 years
3. Grade. 9th, 10th, 11th, or 12th
4. English speaking. Adolescent

Exclusion Criteria:

1. Current diagnosis of substance use or conduct disorder
2. Concurrent mental disorder of greater severity than social anxiety disorder
3. Current psychotic symptoms
4. Current suicidal ideation
5. Pervasive developmental disorder, or a significant medical disorder (e.g., substantially impairs functioning, school attendance, or the ability to engage in treatment)
6. Current psychological or pharmacological treatment

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2010-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in Diagnostic severity of social anxiety disorder (ADIS CSR score) | 2 week and 6-month follow-up
  ADIS CSR Ratings are taken at baseline, immediately following treatment, and at a 6-month followup.
Change in Treatment response/non-response (a CGI-I of Improved or better, ratings of 1-3, 3 = Improved) | 2 week and 6-month follow-up
  CGI-I assesses improvement from baseline immediately following treatment and at a 6-month followup assessment.

SECONDARY OUTCOMES:
Change in Diagnostic status: presence or absence of social anxiety disorder | 2 week and 6-month follow-up
Change in Overall and school functioning: spare-time, peer relations, home life, school attendance, grades, and LSAS-CA school items total score | 2 week and 6-month follow-up
Change in Adolescent and parent ratings of social anxiety scale scores (self and parent SPAI-C), and adolescent ratings of depression (BDI-II) | 2 week and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Masia, Ph.D., Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Masia Warner C, Colognori D, Brice C, Herzig K, Mufson L, Lynch C, Reiss PT, Petkova E, Fox J, Moceri DC, Ryan J, Klein RG. Can school counselors deliver cognitive-behavioral treatment for social anxiety effectively? A randomized controlled trial. J Child Psychol Psychiatry. 2016 Nov;57(11):1229-1238. doi: 10.1111/jcpp.12550. Epub 2016 Mar 22. PMID 27002215